CLINICAL TRIAL: NCT00501514
Title: Effects of Growth Hormone on Exercise Capacity and Cardiopulmonary Performance in Patients With Chronic Heart Failure
Brief Title: Effects of Growth Hormone on Exercise Capacity
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Federico II University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CTN 96-0870-001
Record Dates: First submitted 2007-07-12; First posted 2007-07-16 (Estimated); Last update posted 2009-01-29 (Estimated); Status verified 2009-01

CONDITIONS: Chronic Heart Failure
Keywords: chronic heart failure; cardiopulmonary exercise; oxygen consumption; growth hormone
MeSH Terms: interventions — Growth Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Growth hormone

SUMMARY:
The purpose of this study was to assess whether Growth Hormone(GH)improves exercise capacity and cardiopulmonary performance in patients with chronic heart failure.

DETAILED DESCRIPTION:
clinical studies have focused the effects of GH on left ventricular function and hemodynamics. Little is known about the impact of GH on cardiopulmonary performance and exercise capacity. Such data would be relevant, given the well-recognized importance of cardiopulmonary performance and exercise capacity as markers of disease progression and predictors of mortality in patients with CHF.Consequently we conducted a randomised double blind placebo controlled trial to investigate the effects of a three month course of GH, adjunctive to background therapy, on cardiopulmonary performance and exercise capacity in patients with dilated cardiomyopathy and CHF.The primary outcome of the study was improvement of peak VO2 assessed by a cardiopulmonary exercise testing. Secondary endpoints were exercise capacity and ejection fraction obtained by echocardiography.

ELIGIBILITY:
Inclusion Criteria:

* Ejection fraction < 40%
* Left ventricular internal dimension >58 mm
* II-III NYHA class
* Stable hemodynamic condition during the previous three months
* Sinus rhythm

Exclusion Criteria:

* IMA or CABG or PTCA in the previous six months
* Instable angina
* Major arrhythmias (Lown class> IV)
* Diseases limiting exercise capacity
* Insulin treated diabetes mellitus

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 1997-11; Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
The primary outcome of the study was improvement of peak VO2 assessed by a cardiopulmonary exercise testing. | three months

SECONDARY OUTCOMES:
Secondary endpoints were exercise capacity and ejection fraction obtained by echocardiography. | three months

CONTACTS AND LOCATIONS:
Overall Officials: Luigi Saccà, MD, Principal Investigator — Federico II University
Locations (1):
- Dpt of internal medicine University Federico II, Naples, Italy

REFERENCES:
- [Background] Fazio S, Sabatini D, Capaldo B, Vigorito C, Giordano A, Guida R, Pardo F, Biondi B, Sacca L. A preliminary study of growth hormone in the treatment of dilated cardiomyopathy. N Engl J Med. 1996 Mar 28;334(13):809-14. doi: 10.1056/NEJM199603283341301. PMID 8596546
- [Background] Genth-Zotz S, Zotz R, Geil S, Voigtlander T, Meyer J, Darius H. Recombinant growth hormone therapy in patients with ischemic cardiomyopathy : effects on hemodynamics, left ventricular function, and cardiopulmonary exercise capacity. Circulation. 1999 Jan 5-12;99(1):18-21. doi: 10.1161/01.cir.99.1.18. PMID 9884373
- [Background] Osterziel KJ, Strohm O, Schuler J, Friedrich M, Hanlein D, Willenbrock R, Anker SD, Poole-Wilson PA, Ranke MB, Dietz R. Randomised, double-blind, placebo-controlled trial of human recombinant growth hormone in patients with chronic heart failure due to dilated cardiomyopathy. Lancet. 1998 Apr 25;351(9111):1233-7. doi: 10.1016/S0140-6736(97)11329-0. PMID 9643742